CLINICAL TRIAL: NCT05957172
Title: Mobile Advanced Multi-Parameter Reporting in Patients Wearing a Novel Device: Utilization During Cardiac Rehabilitation
Acronym: MAPS-III
Status: Withdrawn | Type: Observational
Why Stopped: Futility
Sponsor: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 90D0257
Record Dates: First submitted 2023-01-23; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Heart Attack; Cardiac Event; Cardiac Disease; Cardiac Infarct; NSTEMI; STEMI
Keywords: heart attack; myocardial infarction; STEMI; NSTEMI
MeSH Terms: conditions — Myocardial Infarction; Cardiovascular Diseases; Heart Diseases; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Active Treatment: Subjects assigned to wear the FDA-cleared AMS device for 30-60 days Sequential enrollment to avoid preferential selection Investigator blinded to the AMS data
  Interventions: Device: ZOLL Arrhythmia Management System

INTERVENTIONS:
Device: ZOLL Arrhythmia Management System — AMS records rhythm, heart rate, subject-reported symptoms, and multiple parameters that include respiration rate, activity, and body posture (biometric data)
  Other Names: AMS

SUMMARY:
Advanced remote multi-parameter reporting during cardiac rehabilitation (MAPS-III). The primary purpose of this observational study is to collect baseline information of cardiac rehabilitation usage in the US for post-myocardial infarction (MI) patients with EF > 35% while wearing the ZOLL AMS device for 30 to 60 days. Secondary data on biometrics, arrhythmias, symptoms, and healthcare utilization will provide additional background information on this population during the early post-MI cardiac rehabilitation period.

DETAILED DESCRIPTION:
To collect baseline data on cardiac rehabilitation usage (referrals and completion) in recent post-MI patients with EF > 35%.To collect data on AMS-derived biometric data (e.g. HR, activity) and arrhythmias, and subject-reported symptoms, beta blocker/ivabradine usage (dose/changes) and cardiovascular events. The participating centers will enroll consenting subjects in a sequential manner to avoid preferential selection of patients to participate in the study. Subjects will be consented by the center study staff, and if eligible will wear the FDA-cleared AMS device for 30-60 days. Subject demographic information and clinical history will be obtained at the time of enrollment. During the study period, the prescribing physician-investigator will be blinded to AMS data. Final subject follow-up will be at 3 months. A sample size of 150 subjects is estimated in order to have 100 subjects with at least 30 days of AMS use for analysis.

ELIGIBILITY:
Inclusion Criteria

1. Both male and female subjects who are between 21 - 75 years of age, inclusively
2. Subjects who are consented and enrolled into the study prior to discharge from the qualifying acute myocardial infarction
3. Subjects with a consistent EF >35% post the qualifying acute myocardial infarction

Exclusion Criteria

1. Subjects with an implantable cardiac device such as left ventricular assistive device, pacemaker, an implanted cardioverter defibrillator (ICD), a cardiac resynchronization therapy device, subcutaneous ICDs, pressure monitors, and loop monitors.
2. Subjects with wearable cardioverter defibrillator, Holter monitors, wearable event recorders, and other mobile cardiac telemetry devices at the same time.
3. Subjects with a skin condition preventing them from wearing the AMS device.
4. Subjects who are non-ambulatory for any reason.
5. Subjects who are self-reporting to be pregnant.
6. Subjects with comorbidities that would preclude adherence to a cardiac rehabilitation program - at the discretion of the physician.
7. Subjects participating or planning to participate in another interventional study during the protocol-defined study period

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post-MI patients with an EF >35% undergoing cardiac rehabilitation
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Cardiac rehabilitation program referrals and completions (in-clinic or home-based) | 30-60 days
  Measure the completion rate of patients undergoing cardiac rehabilitation programs i.e. the number of cardiac rehabilitation program referrals vs. number of cardiac rehabilitation program completions

SECONDARY OUTCOMES:
AMS-derived data - Heart Rate | 30-60 days
  Improvement in nighttime resting heart rate
AMS-derived data - Activity | 30-60 days
  Changes in total daily activity as detected by the AMS accelerometers
AMS-derived data - Arrhythmias | 30-60 days
  Occurrence of Arrhythmias as detected by the AMS
Subject reported outcomes - Beta blocker/ivabradine usage/changes | 30-60 days
  Initiation/Termination/Changes in beta blocker/ivabradine usage recorded via weekly diary
Subject reported outcomes - Symptoms | 30-60 days
  Occurrence and changes in symptoms recorded via weekly diary
Subject reported outcomes - Cardiovascular events | 30-60 days
  Cardiovascular events as measured by health care use i.e. unplanned health care provider visits due to cardiovascular event, recorded via weekly diary